CLINICAL TRIAL: NCT01872130
Title: Reflectance Confocal Microscopy of Wounds During Moh's Surgery: Feasibility Testing of a Mosaicing Algorithm for Intraoperative Imaging of Cancer Margins
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12-239
Record Dates: First submitted 2013-05-31; First posted 2013-06-07 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma
Keywords: Moh's Surgery; mosaicing algorithm; intraoperative imaging; 12-239
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate a new instrument that shines light and takes digital pictures of skin. The goal is to develop a technique that may enable fast and accurate assessment of surgical margins in the excision of basal cell carcinoma (BCC) or squamous cell carcinoma (SCC). The investigators will evaluate the pictures obtained by the confocal microscope to determine whether this technique may be useful in the future for helping Mohs surgeons remove cancers. In the future, patients may benefit with shorter surgery and improved care.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Mohs surgery for basal cell carcinoma (BCC )or squamous cell carcinoma (SCC). .
* Ability to sign informed consent.
* Age ≥ 18 years.

Exclusion Criteria:

* Mohs surgery located on a site that may not be convenient to confocal imaging.
* Inability to give informed consent.
* Inability to tolerate imaging procedure (i.e., remain relatively still for multiple short durations of 3-4 minutes) over a total time of 20 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Dermatology clinics at MSKCC
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-05; Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
test feasibility of a mosaicing algorithm intraoperative | 1 year
  For the primary study objective, the Mohs surgeon will perform a qualitative assessment of the confocal mosaic. This will be a dichotomous assessment of whether the mosaic is of sufficient quality (contrast and resolution) to identify individual features. The specific features for BCC or SCC margins are tumor nests with nuclear atypia and increased nuclear density (relative to the density seen in normal basal cells).

SECONDARY OUTCOMES:
test feasibility of a mosaicing algorithm preoperative | 1 year
  imaging of cancer margins on patients, before Mohs surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Kishwer Nehal, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center Hauppauge, Hauppauge, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/